CLINICAL TRIAL: NCT00331604
Title: Inhaled Pre-prandial Human Insulin With the AERx® iDMS Versus s.c. Insulin Aspart in Type 2 Diabetes: A 104 Week, Open-label, Multicenter, Randomised, Trial Followed by a 12 Week Re-randomised Extension to Investigate Safety and Efficacy
Brief Title: Safety and Efficacy of Inhaled Insulin in Type 2 Diabetes
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: See termination reason in detailed description
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN1998-2161; 2005-005378-58 (EudraCT Number)
Record Dates: First submitted 2006-05-24; First posted 2006-05-31 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental)
  Interventions: Drug: inhaled human insulin; Drug: insulin detemir
- B (Active Comparator)
  Interventions: Drug: insulin detemir; Drug: insulin aspart
- C (Active Comparator)
  Interventions: Drug: insulin detemir; Drug: insulin aspart

INTERVENTIONS:
Drug: inhaled human insulin — Treat-to-target dose titration scheme, inhalation.
  Arms: A
Drug: insulin detemir — Injection s.c., 50% of daily dose.
  Other Names: NN304; Levemir
Drug: insulin aspart — Treat-to-target dose titration scheme, injection s.c.
  Arms: B; C
Drug: insulin aspart — Treat-to-target dose titration scheme, injection s.c. After 2 years.
  Arms: C

SUMMARY:
This trial is conducted in Asia, Europe and South America. The aim of this research is to compare the efficacy (reduction in HbA1c and blood glucose) and pulmonary safety (pulmonary function tests, chest x-rays) of mealtime inhaled insulin with subcutaneous insulin aspart both in combination with insulin detemir in Type 2 Diabetes.

DETAILED DESCRIPTION:
The decision to discontinue the development of AERx® is not due to any safety concerns. An analysis concluded that fast-acting inhaled insulin in the form it is known today, is unlikely to offer significant clinical or convenience benefits over injections of modern insulin with pen devices.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Currently treated with insulin
* Body mass index of (BMI) less than or equal to 40.0 kg/m2
* HbA1c less than or equal to 11.0%

Exclusion Criteria:

* Total daily insulin dosage less than or equal to 100 IU or U/day
* Current smoking or smoking within the last 6 months
* Cardiac problems
* Uncontrolled hypertension
* Current proliferative retinopathy or maculopathy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 618 (Actual)
Dates: Start 2006-08-31 (Actual); Primary Completion 2008-05-05 (Actual); Study Completion 2008-05-05 (Actual)

PRIMARY OUTCOMES:
Treatment difference in HbA1c | After 52 weeks

SECONDARY OUTCOMES:
Adverse events | For the duration of the trial
Blood glucose | After 52, 104 and 116 weeks of treatment
Body weight | During treatment
Lung function | After 52, 104 and 116 weeks of treatment
Hypoglycaemia | From 12 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (68):
- Brazil (4):
  - Novo Nordisk Investigational Site, Campinas
  - Novo Nordisk Investigational Site, Higienópolis
  - Novo Nordisk Investigational Site, Porto Alegre
  - Novo Nordisk Investigational Site, São Paulo
- Denmark (3):
  - Novo Nordisk Investigational Site, Århus C
  - Novo Nordisk Investigational Site, Hillerød
  - Novo Nordisk Investigational Site, Hvidovre
- France (8):
  - Novo Nordisk Investigational Site, Brest
  - Novo Nordisk Investigational Site, Grenoble
  - Novo Nordisk Investigational Site, La Rochelle
  - Novo Nordisk Investigational Site, Nanterre
  - Novo Nordisk Investigational Site, Narbonne
  - Novo Nordisk Investigational Site, Nevers
  - Novo Nordisk Investigational Site, Strasbourg
  - Novo Nordisk Investigational Site, Toulouse
- Germany (15):
  - Novo Nordisk Investigational Site, Bad Harzburg
  - Novo Nordisk Investigational Site, Bad Kreuznach
  - Novo Nordisk Investigational Site, Bad Lauterberg im Harz
  - Novo Nordisk Investigational Site, Dresden
  - Novo Nordisk Investigational Site, Friedrichsthal
  - Novo Nordisk Investigational Site, Hamburg
  - Novo Nordisk Investigational Site, Herrenberg
  - Novo Nordisk Investigational Site, Hohenmölsen
  - Novo Nordisk Investigational Site, Neumünster
  - Novo Nordisk Investigational Site, Neuwied
  - Novo Nordisk Investigational Site, Saint Ingbert
  - Novo Nordisk Investigational Site, Schkeuditz
  - Novo Nordisk Investigational Site, Speyer
  - Novo Nordisk Investigational Site, Völklingen
  - Novo Nordisk Investigational Site, Warburg
- Novo Nordisk Investigational Site, Shatin, New Territories, Hong Kong
- Israel (3):
  - Novo Nordisk Investigational Site, Beersheba
  - Novo Nordisk Investigational Site, Holon
  - Novo Nordisk Investigational Site, Jerusalem
- Italy (10):
  - Novo Nordisk Investigational Site, Bari
  - Novo Nordisk Investigational Site, Catania
  - Novo Nordisk Investigational Site, Catanzaro
  - Novo Nordisk Investigational Site, Milan
  - Novo Nordisk Investigational Site, Perugia
  - Novo Nordisk Investigational Site, Pescara
  - Novo Nordisk Investigational Site, Pisa
  - Novo Nordisk Investigational Site, Roma
  - Novo Nordisk Investigational Site, San Giovanni Rotondo
  - Novo Nordisk Investigational Site, Verona
- Novo Nordisk Investigational Site, Singapore, Singapore
- Spain (9):
  - Novo Nordisk Investigational Site, Almería
  - Novo Nordisk Investigational Site, Cáceres
  - Novo Nordisk Investigational Site, Elche
  - Novo Nordisk Investigational Site, Granada
  - Novo Nordisk Investigational Site, Lugo
  - Novo Nordisk Investigational Site, Mostoles - Madrid -
  - Novo Nordisk Investigational Site, Seville
  - Novo Nordisk Investigational Site, Valladolid
  - Novo Nordisk Investigational Site, Xátiva
- Taiwan (2):
  - Novo Nordisk Investigational Site, Taichung
  - Novo Nordisk Investigational Site, Taipei
- United Kingdom (12):
  - Novo Nordisk Investigational Site, Aberdeen
  - Novo Nordisk Investigational Site, Ayr
  - Novo Nordisk Investigational Site, Bristol
  - Novo Nordisk Investigational Site, Cosham
  - Novo Nordisk Investigational Site, Edgbaston, Birmingham
  - Novo Nordisk Investigational Site, Edinburgh
  - Novo Nordisk Investigational Site, Livingstone
  - Novo Nordisk Investigational Site, Nottingham
  - Novo Nordisk Investigational Site, Plymouth
  - Novo Nordisk Investigational Site, Salford
  - Novo Nordisk Investigational Site, Sheffield
  - Novo Nordisk Investigational Site, Wirral, Merseyside

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com